CLINICAL TRIAL: NCT05758233
Title: Comparison of the Effectiveness of Ultrasound-guided Transversalis Fascia Plane Block and Transversus Abdominis Plane Block on Postoperative Pain in Caesarean Section : a Prospective Randomized Trial
Brief Title: The Effect of Peripheral Nerve Blocks on Postoperative Analgesia in Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-74
Record Dates: First submitted 2023-02-20; First posted 2023-03-07 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia; Sexual; Analgesia
Keywords: anesthesia recovery period; cesarean section; obstetric anesthesia; spinal anaesthesia; postoperative analgesia
MeSH Terms: conditions — Coitus; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective randomize study
Masking Description: prospective randomize study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup 1: Transversalis Fascia Plane Block (TFPB) (Experimental): Transversalis Fascia Plane Block (TFPB)
  Interventions: Procedure: Patients undergoing transversalis fascia plane block; Procedure: Patients undergoing transversus abdominis plane block
- Grup 2: Transversus Abdominis Plane Block (TAPB) (Experimental): Transversus Abdominis Plane Block (TAPB)
  Interventions: Procedure: Patients undergoing transversalis fascia plane block; Procedure: Patients undergoing transversus abdominis plane block

INTERVENTIONS:
Procedure: Patients undergoing transversalis fascia plane block — The investigators applied a transversalis fascia plane block to the group of patients who had a cesarean section under spinal anesthesia to prevent postoperative pain.
Procedure: Patients undergoing transversus abdominis plane block — The investigators applied a transversus abdominis plane block to the group of patients who had a cesarean section under spinal anesthesia to prevent postoperative pain.

SUMMARY:
The goal of this prospective randomized study was to compare the efficacy of transversus abdominis plane block and transversalis fascia plane block for postoperative analgesia in patients undergoing elective cesarean section under spinal anesthesia.

The main question[s] it aims to answer are:

[Is transversalis fascia plane block more effective in postoperative analgesia? ]

[Is there a difference between the duration of postoperative first analgesia requirement? ] Since the pain scores after the block at the end of the operation will be evaluated during the postoperative 24 hours, the participants will be asked to give a value between 0 and 10 in certain time periods.

DETAILED DESCRIPTION:
This prospective, randomized trial was conducted at Başakşehir Çam and Sakura City Hospital by the Declaration of Helsinki. After ethics committee approval (decision no: 2022-74, date: 09.03.2022) and written informed consent was obtained from all patients, the trial was conduct-ed according to Consolidated Standards of Reporting Trials (CONSORT) guidelines.A total of 150 patients were divided into two groups: transversal fascia plane block (TFPB group) and Transversus abdominis plane block (TAPB group).VAS values, time to first analgesic requirement, analgesic requirements, nausea & vomiting and pruritus were evaluated for 24 hours postoperatively (6th hour (T2), 12th hour (T3), 24th hour .

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years old pregnant woman
* ASAII-III
* Patients accepting spinal anesthesia

Exclusion Criteria:

* Morbid obesity(BMI >40)
* Patients who are switched to general anesthesia in an unexpected perioperative situation
* Patients with placental anomaly
* Patients with bupivacaine allergy
* Fetal distress situations too urgent to wait for spinal anesthesia and patients who do not want spinal anesthesia

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 20-50 age
Enrollment: 150 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
time of first analgesic need | 24 hours postoperatively
  Our primary goal was to meet the initial analgesic requirement times.

SECONDARY OUTCOMES:
visuel analog scale | 24 hours postoperatively
  Our secondary aim was to compare postoperative pain scores. The first 24 hours postoperatively were evaluated.Visual analog scale(VAS) was used to assess postoperative pain.6th, 12th, 24th hour VAS values were recorded For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akyol, M.D, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryu C, Choi GJ, Jung YH, Baek CW, Cho CK, Kang H. Postoperative Analgesic Effectiveness of Peripheral Nerve Blocks in Cesarean Delivery: A Systematic Review and Network Meta-Analysis. J Pers Med. 2022 Apr 14;12(4):634. doi: 10.3390/jpm12040634. PMID 35455750
- [Result] Mitchell KD, Smith CT, Mechling C, Wessel CB, Orebaugh S, Lim G. A review of peripheral nerve blocks for cesarean delivery analgesia. Reg Anesth Pain Med. 2019 Oct 25:rapm-2019-100752. doi: 10.1136/rapm-2019-100752. Online ahead of print. PMID 31653797